CLINICAL TRIAL: NCT04742491
Title: HPTN 091: Integrating HIV Prevention, Gender-Affirmative Medical Care, and Peer Health Navigation for Transgender Women in the Americas: A Vanguard Study
Brief Title: Pre-Exposure Prophylaxis for Transgender Women in the US and South America
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 091
Record Dates: First submitted 2020-11-30; First posted 2021-02-08 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention
Keywords: Transgender women; TGW
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Intermediate Intervention Arm vs. Deferred Intervention Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immediate Intervention Arm (Experimental): PrEP (pre-exposure prophylaxis) provision, STI screening and treatment, GAHT (gender-affirming hormonal therapy), peer-health management using strengths-based management. PrEP provision includes using one daily tablet of Descovy (emtricitabine 200 mg and tenofovir alafenamide 25mg, FTC/TAF) or one daily tablet of Truvada (emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg, FTC/TDF) in the US, and one daily tablet of Truvada (emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg, FTC/TDF) in Brazil.
  Interventions: Drug: Immediate Intervention Arm
- Deferred Intervention Arm (Experimental): 0-6 months PrEP (pre-exposure prophylaxis) provision and STI screening and treatment. From months 6-18, GAHT (gender-affirming hormonal therapy) and peer-health management using strengths-based management. PrEP provision includes one daily tablet of Descovy (emtricitabine 200 mg and tenofovir alafenamide 25mg, FTC/TAF) or one daily tablet of Truvada (emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg, FTC/TDF) in the US, and one daily table of Truvada (emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg, FTC/TDF) in Brazil.
  Interventions: Drug: Deferred Intervention Arm

INTERVENTIONS:
Drug: Immediate Intervention Arm — Truvada, Descovy in the United States; Truvada in Brazil
  Other Names: Truvada, Descovy
  Arms: Immediate Intervention Arm
Drug: Deferred Intervention Arm — Truvada, Descovy in the United States; Truvada in Brazil
  Other Names: Truvada, Descovy
  Arms: Deferred Intervention Arm

SUMMARY:
A study to assess the feasibility, acceptability, and preliminary impact of a multi-component strategy to improve pre-exposure prophylaxis (PrEP) uptake and adherence that integrates delivery of biomedical HIV prevention co-located with gender-affirming transgender care (hormonal therapy and medical monitoring) and Peer Health Navigation (PHN) using Strengths-Based Case Management (SBCM) professional supervision.

Multi-site, open-label study with each participant randomized 1:1 to Immediate Intervention vs. 6-month Deferred Intervention Arms. Both arms will be provided PrEP and sexually transmitted infection (STI) screening and treatment. Participants in the Immediate Intervention Arm will receive co-located gender-affirming medical care and PHN using SBCM starting at the Enrollment Visit. Participants in the Deferred Intervention Arm will receive linkage to external gender-affirming medical care and case management services during the deferred period and will transition to the study intervention six months following the Enrollment Visit.

DETAILED DESCRIPTION:
entered elsewhere

ELIGIBILITY:
Inclusion Criteria:

* TGW (assigned male at birth, trans-feminine spectrum - as defined in the SSP Manual - by self-report) who meet all of the following criteria are eligible for inclusion in this study.
* Eighteen years or older at the time of screening.
* Willing and able to provide informed consent for the study.
* Interest in PrEP - as defined in the SSP Manual.
* Non-reactive HIV test results at Screening and Enrollment.
* Available to return for all study visits and within site catchment area, as defined per site's Standard Operating Procedures (SOP).
* At risk for sexually acquiring HIV infection based on self-report of at least one of the following:

  1. Any anal or vaginal sex with one or more serodiscordant or HIV-unknown serostatus sexual partners in the previous 3 months, regardless of condom use.
  2. Anal or vaginal sex in exchange for money, food, shelter, or other goods or favors in the previous 3 months.
  3. History of STI(s) in the past 6 months.
* Willing to undergo all required study procedures.
* General good health, as evidenced by the following laboratory values:

  1. Calculated creatinine clearance ≥ 60 mL/minute using the Cockcroft-Gault equation.
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 times the upper limit of normal (ULN.)
  3. HBV surface antigen (HBsAg) negative.

Note: Otherwise eligible participants with laboratory results outside the above-mentioned values, with the exception of those with reactive HIV test, can be re-tested during the screening window. Participants with reactive HIV tests will not be able to rescreen.

Note: Participants who practice receptive vaginal sex cannot be provided Descovy® as it is not approved for this indication.

Exclusion Criteria:

1. Any reactive or positive HIV test result at Screening or Enrollment, even if HIV infection is not confirmed.
2. Plans to move away from the site area within the next 18 months.
3. Co-enrollment in any other research study that may interfere with this study (as provided by self-report or other available documentation). Exceptions may be made after consultation with the Clinical Management Committee (CMC).
4. Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy).
5. History of deep vein thrombosis, pulmonary embolism, and/or clotting disorder.
6. Active or planned use of medications with significant drug interactions as described in the Package Insert for Truvada® or Descovy®, per clinician's discretion (provided by selfreport or obtained from medical history or medical records). See Section 5.8 for a full list of drug interactions.
7. Any other condition, including but not limited to alcohol or substance abuse and uncontrolled medical condition and/or allergies, that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives would make the patient unsuitable for the study or unable/unwilling to comply with the study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender Women
Enrollment: 304 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonia Poteat, PhD, MPH, Study Chair — UNC Chapel Hill
Locations (5):
- United States (4):
  - Bridge HIV CRS, San Francisco, California
  - Harlem Prevention Center CRS, New York, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas
- Instituto de Pesquisa Clinicaq Evandro Chagas CRS, Manguinhos, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were randomized to study arms.
Groups:
- Immediate Intervention Arm: PrEP, GAHT and peer-health management was provided from enrollment to study exit.
- Deferred Intervention Arm: PrEP was provided from enrollment to study exit.
  GAHT and peer-health management were offered from month 6 (week 26) to study exit.
Period: Overall Study
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Started | 149 | 155
Week 13 Follow-up | 133 | 139
Week 26 Follow-up | 125 | 136
Week 39 Follow-up | 118 | 128
Week 52 Follow-up | 116 | 123
Week 65 Follow-up | 114 | 126
Completed | 126 | 128
Not Completed | 23 | 27
Not completed — Death | 2 | 0
Not completed — Participant unwilling or unable to comply with required study procedures | 1 | 1
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 4 | 2
Not completed — One or more reactive HIV test results or acute HIV infection suspected | 2 | 1
Not completed — Participant refused further participation | 2 | 7
Not completed — Participant unable to adhere to visit schedule | 3 | 4
Not completed — Other reasons | 3 | 4

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the assignment in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm | Total
Number analyzed (Participants) | 149 | 155 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.8) | 30.9 (8.8) | 30.6 (8.8)
Age, Customized [Count of Participants; unit: Participants] — Age (in years) dichotomized as 25 and below, and 26 and above.
  Participants
    25 and below | 57 | 47 | 104
    26 and above | 92 | 108 | 200
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Missing | 0 | 1 | 1
  Gender: Female | 28 | 20 | 48
  Gender: Transgender Female/Transgender Woman | 65 | 76 | 141
  Gender: Gender nonbinary/Genderfluid/Gender Nonconforming | 3 | 9 | 12
  Gender: Another gender identity | 4 | 5 | 9
  Gender: Prefer not to answer | 0 | 0 | 0
  Gender: Multiple gender identities selected | 49 | 44 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 149 | 155 | 304
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 82 | 81 | 163
  Not Hispanic or Latino | 62 | 72 | 134
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 46 | 50 | 96
  White | 53 | 54 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: PrEP Uptake
Description: Time to PrEP initiation is defined as the duration from enrollment to the PrEP start date.
Time Frame: 0-18 months
Population: Limited to participants who obtained PrEP at the study clinic
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
days | 16.2 (66.7) | 11.4 (4.3)

2. Primary Outcome: PrEP Adherence
Description: Self-reported adherence to daily PrEP by study visit
Time Frame: 0-18 months
Population: Number of participants who completed CASI at each study visit. Due to missingness, this number may be lower than the number of participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment: < 2 doses per week | 2 | 1
  Enrollment: 2-3 doses per week | 2 | 3
  Enrollment: 4-6 doses per week | 6 | 4
  Enrollment: 7 doses per week | 19 | 20
  Enrollment: Missing | 118 | 125
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13: < 2 doses per week | 3 | 8
  Week 13: 2-3 doses per week | 2 | 3
  Week 13: 4-6 doses per week | 19 | 27
  Week 13: 7 doses per week | 79 | 75
  Week 13: Missing | 30 | 26
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26: < 2 doses per week | 7 | 7
  Week 26: 2-3 doses per week | 7 | 2
  Week 26: 4-6 doses per week | 12 | 21
  Week 26: 7 doses per week | 76 | 72
  Week 26: Missing | 22 | 29
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39: < 2 doses per week | 4 | 4
  Week 39: 2-3 doses per week | 3 | 5
  Week 39: 4-6 doses per week | 16 | 23
  Week 39: 7 doses per week | 61 | 71
  Week 39: Missing | 30 | 25
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52: < 2 doses per week | 4 | 5
  Week 52: 2-3 doses per week | 3 | 5
  Week 52: 4-6 doses per week | 18 | 16
  Week 52: 7 doses per week | 53 | 63
  Week 52: Missing | 37 | 31
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65: < 2 doses per week | 2 | 5
  Week 65: 2-3 doses per week | 1 | 5
  Week 65: 4-6 doses per week | 16 | 21
  Week 65: 7 doses per week | 57 | 61
  Week 65: Missing | 33 | 30
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78: < 2 doses per week | 3 | 9
  Week 78: 2-3 doses per week | 7 | 7
  Week 78: 4-6 doses per week | 17 | 16
  Week 78: 7 doses per week | 51 | 61
  Week 78: Missing | 47 | 36

3. Primary Outcome: Acceptability and Feasibility of Co-located Services
Description: Number of participants accepting co-located GAHT services at baseline and subsequent quarterly study visits.
Time Frame: 0-18 months
Population: Enrolled participants. Deferred arm participants receive co-located services at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment | 68 | 0
  Week 13 | 106 | 0
  Week 26 | 109 | 66
  Week 39 | 113 | 90
  Week 52 | 114 | 93
  Week 65 | 115 | 93
  Week 78 | 116 | 93

4. Primary Outcome: Participant Retention at Weeks 26, 52 and 78
Description: Participant retention at weeks 26, 52 and 78 by study arm. Retention defined as the number of participants who completed the visit divided by the number of participants who are expected or have completed the visit.
Time Frame: Weeks 26, 52, 78
Population: The denominators in the table differ from the overall number analyzed because the denominator excludes any participants who have terminated from the study or seroconverted at the time of the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Week 26: number analyzed (Participants) | 147 | 151
  Week 26 | 125 | 135
  Week 52: number analyzed (Participants) | 140 | 144
  Week 52 | 115 | 123
  Week 78: number analyzed (Participants) | 136 | 143
  Week 78 | 126 | 128

5. Primary Outcome: Acceptability and Feasibility of Peer Health Navigation
Description: The average number of peer health navigator encounters.
Time Frame: 0-18 months
Population: Enrolled population
Measure: Mean (Standard Deviation); unit: encounters
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
encounters | 5.7 (1.6) | 5.5 (1.2)

6. Primary Outcome: Acceptability and Feasibility of Peer Health Navigation
Description: Number of each type of peer health navigation encounter.
Time Frame: 0-18 months
Population: Total number of peer health navigation encounters by arm.
Measure: Count of Units; unit: Encounters
Units Other Than Participants: Encounters
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Number analyzed (Encounters) | 839 | 737
Encounters
  In-person | 519 | 427
  Email | 0 | 0
  Text | 16 | 7
  Phone | 258 | 256
  Video encounter | 46 | 47

7. Primary Outcome: Acceptability and Feasibility of Co-located Services
Description: Percentage of participants who report desire for co-located services at the end of the study
Time Frame: 0-18 months
Population: Participants with a non-missing response to the CASI question concerning desire for co-located services at the end of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 145 | 149
Participants | 106 | 107
Statistical Analysis 1: Comparison: Immediate Intervention Arm; Test type: Superiority; p = 0.80, Chi-squared; Percentage = 73.10, 95% CI 2-sided [65.89 to 80.30]; The estimates and C.I. (In percentage) are derived using Chi-squared test
Statistical Analysis 2: Comparison: Deferred Intervention Arm; Test type: Superiority; p = 0.80, Chi-squared; Percentage = 71.81, 95% CI 2-sided [64.59 to 79.04] — The estimates and C.I. (In percentage) are derived using Chi-squared test

8. Primary Outcome: PrEP Adherence
Description: The average number of days to first PrEP permanent discontinuation.
Time Frame: 0-18 months
Population: Participants who initiated PrEP and had at least one permanent discontinuation prior to study exit or termination.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 28 | 18
days | 364.1 (185.2) | 361.1 (255.2)

9. Primary Outcome: PrEP Adherence
Description: The median number of days to first PrEP permanent discontinuation.
Time Frame: 0-18 months
Population: Participants who initiated PrEP and had at least one permanent discontinuation prior to study exit or termination.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 28 | 18
days | 373 [245 to 499] | 409 [141 to 533]

10. Primary Outcome: PrEP Adherence
Description: Participants with different levels of TFV-DP concentrations in DBS measured at quarterly follow-up visits after PrEP initiation.
Time Frame: 0-18 months
Population: TFVDP levels of participants who obtained PrEP at the study clinic.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
Participants
  Enrollment: number analyzed (Participants) | 105 | 117
  Enrollment: Unquantifiable | 80 | 83
  Enrollment: Less than 2 doses per week | 10 | 15
  Enrollment: 2-3 doses per week | 5 | 3
  Enrollment: 4-6 doses per week | 5 | 12
  Enrollment: 7 doses per week | 5 | 4
  Week 13: number analyzed (Participants) | 111 | 115
  Week 13: Unquantifiable | 19 | 10
  Week 13: Less than 2 doses per week | 23 | 25
  Week 13: 2-3 doses per week | 6 | 10
  Week 13: 4-6 doses per week | 28 | 27
  Week 13: 7 doses per week | 35 | 43
  Week 26: number analyzed (Participants) | 108 | 120
  Week 26: Unquantifiable | 21 | 20
  Week 26: Less than 2 doses per week | 23 | 28
  Week 26: 2-3 doses per week | 8 | 12
  Week 26: 4-6 doses per week | 32 | 26
  Week 26: 7 doses per week | 24 | 34
  Week 39: number analyzed (Participants) | 100 | 112
  Week 39: Unquantifiable | 31 | 23
  Week 39: Less than 2 doses per week | 19 | 19
  Week 39: 2-3 doses per week | 6 | 9
  Week 39: 4-6 doses per week | 22 | 27
  Week 39: 7 doses per week | 22 | 34
  Week 52: number analyzed (Participants) | 100 | 110
  Week 52: Unquantifiable | 29 | 22
  Week 52: Less than 2 doses per week | 18 | 17
  Week 52: 2-3 doses per week | 14 | 8
  Week 52: 4-6 doses per week | 19 | 32
  Week 52: 7 doses per week | 20 | 31
  Week 65: number analyzed (Participants) | 98 | 113
  Week 65: Unquantifiable | 27 | 21
  Week 65: Less than 2 doses per week | 19 | 26
  Week 65: 2-3 doses per week | 12 | 9
  Week 65: 4-6 doses per week | 17 | 22
  Week 65: 7 doses per week | 23 | 35
  Week 78: number analyzed (Participants) | 110 | 114
  Week 78: Unquantifiable | 39 | 32
  Week 78: Less than 2 doses per week | 22 | 20
  Week 78: 2-3 doses per week | 10 | 12
  Week 78: 4-6 doses per week | 16 | 23
  Week 78: 7 doses per week | 23 | 27

11. Primary Outcome: PrEP Adherence
Description: Participants with different levels FTC-TP concentrations in DBS measured at quarterly follow-up visits after PrEP initiation.
Time Frame: 0-18 months
Population: FTC-TP levels of participants who obtained PrEP at the study clinic.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
Participants
  Enrollment: number analyzed (Participants) | 105 | 117
  Enrollment | 15 | 20
  Week 13: number analyzed (Participants) | 111 | 115
  Week 13 | 73 | 87
  Week 26: number analyzed (Participants) | 108 | 120
  Week 26 | 67 | 74
  Week 39: number analyzed (Participants) | 100 | 112
  Week 39 | 51 | 75
  Week 52: number analyzed (Participants) | 100 | 110
  Week 52 | 52 | 75
  Week 65: number analyzed (Participants) | 98 | 113
  Week 65 | 55 | 70
  Week 78: number analyzed (Participants) | 110 | 114
  Week 78 | 51 | 59

12. Primary Outcome: PrEP Adherence
Description: The proportion of TGW determined to be adherent at the Week 26 visit was compared by study arm. PrEP adherence was defined as having a detectable concentration of PrEP (Truvada or Descovy) in DBS sample.
Time Frame: Week 26
Population: Participants who obtained PrEP at the study clinic.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 108 | 120
Participants | 87 | 100
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Test type: Superiority; p = 0.59, Binomial Distribution

13. Primary Outcome: PrEP Persistent
Description: PrEP persistent is defined as the proportion of study visits where a participant demonstrates high adherence to PrEP among those who initiated PrEP at the study clinic. High adherence at a visit is based on drug concentrations in dried blood spots (DBS):
  Truvada (TDF/FTC): TFV-DP ≥ 900 fmol/punch Descovy (TAF/FTC): TFV-DP ≥ 950 fmol/punch PrEP persistent reflects sustained high PrEP adherence across multiple visits over time, rather than high PrEP adherence at a single point.
Time Frame: 0-18 months
Population: Participants who obtained PrEP at the study clinic.
Measure: Mean (Standard Deviation); unit: percent of visits
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
percent of visits | 41.7 (40.9) | 50.5 (43.2)

14. Primary Outcome: PrEP Uptake
Description: Comparison of PrEP uptake between study arms at the end of Week 26. PrEP uptake is defined as whether the participant initiated PrEP at the study clinic..
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants | 127 | 135
Statistical Analysis 1: Comparison: Immediate Intervention Arm; Test type: Other; p = 0.6381, Binomial Distribution; Percentage = 85.23, 95% CI 2-sided [79.54 to 90.93] — The estimates and C.I. (In percentage) are derived using binomial distribution
Statistical Analysis 2: Comparison: Deferred Intervention Arm; Test type: Other; p = 0.6381, Binomial Distribution; Percentage = 87.10, 95% CI 2-sided [81.82 to 92.37] — The estimates and C.I. (In percentage) are derived using binomial distribution

15. Secondary Outcome: Examining Changes in Sexual Risk-taking Behavior
Description: Describing condom use with HIV+ people, measured by assessments at enrollment and quarterly through Week 78.
Time Frame: 0-18 months
Population: The numbers presented in "Overall Number of Participants Analyzed" represent the total number of participants enrolled in the study. For each visit (row), only participants who completed the CASI questionnaire were included in the analysis. For both questions "condom use with HIV+ people" and "condom use with HIV unknown people" analyses were restricted to participants who completed the CASI questionnaire at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment: Missing | 0 | 1
  Enrollment: No sex | 9 | 12
  Enrollment: Oral sex only | 10 | 7
  Enrollment: I did not have sex with anyone whom I knew was HIV+ | 101 | 88
  Enrollment: None of the time | 11 | 19
  Enrollment: Less than half the time | 3 | 7
  Enrollment: About half the time | 2 | 4
  Enrollment: More than half the time | 5 | 4
  Enrollment: All of the time | 6 | 11
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13: Missing | 0 | 1
  Week 13: No sex | 11 | 16
  Week 13: Oral sex only | 10 | 8
  Week 13: I did not have sex with anyone whom I knew was HIV+ | 81 | 87
  Week 13: None of the time | 7 | 8
  Week 13: Less than half the time | 6 | 3
  Week 13: About half the time | 1 | 3
  Week 13: More than half the time | 9 | 1
  Week 13: All of the time | 8 | 12
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26: Missing | 0 | 1
  Week 26: No sex | 18 | 14
  Week 26: Oral sex only | 17 | 9
  Week 26: I did not have sex with anyone whom I knew was HIV+ | 69 | 80
  Week 26: None of the time | 6 | 8
  Week 26: Less than half the time | 3 | 6
  Week 26: About half the time | 3 | 1
  Week 26: More than half the time | 1 | 3
  Week 26: All of the time | 7 | 9
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39: Missing | 0 | 2
  Week 39: No sex | 13 | 13
  Week 39: Oral sex only | 13 | 9
  Week 39: I did not have sex with anyone whom I knew was HIV+ | 68 | 75
  Week 39: None of the time | 6 | 12
  Week 39: Less than half the time | 3 | 3
  Week 39: About half the time | 2 | 3
  Week 39: More than half the time | 4 | 3
  Week 39: All of the time | 5 | 8
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52: Missing | 4 | 6
  Week 52: No sex | 18 | 12
  Week 52: Oral sex only | 2 | 9
  Week 52: I did not have sex with anyone whom I knew was HIV+ | 65 | 67
  Week 52: None of the time | 7 | 12
  Week 52: Less than half the time | 4 | 5
  Week 52: About half the time | 1 | 2
  Week 52: More than half the time | 5 | 1
  Week 52: All of the time | 9 | 6
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65: Missing | 4 | 7
  Week 65: No sex | 16 | 18
  Week 65: Oral sex only | 6 | 2
  Week 65: I did not have sex with anyone whom I knew was HIV+ | 62 | 70
  Week 65: None of the time | 5 | 9
  Week 65: Less than half the time | 4 | 3
  Week 65: About half the time | 2 | 1
  Week 65: More than half the time | 3 | 0
  Week 65: All of the time | 7 | 12
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78: Missing | 9 | 4
  Week 78: No sex | 23 | 20
  Week 78: Oral sex only | 2 | 0
  Week 78: I did not have sex with anyone whom I knew was HIV+ | 70 | 79
  Week 78: None of the time | 4 | 12
  Week 78: Less than half the time | 3 | 3
  Week 78: About half the time | 6 | 1
  Week 78: More than half the time | 1 | 2
  Week 78: All of the time | 7 | 8

16. Secondary Outcome: Examining Changes in Sexual Risk-taking Behavior
Description: Describing condom use with HIV unknown people, measured by assessments at enrollment and quarterly through Week 78.
Time Frame: 0-18 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment: Missing | 0 | 1
  Enrollment: No sex | 9 | 12
  Enrollment: Oral sex only | 10 | 7
  Enrollment: No sex with anyone whose HIV status was unknown | 30 | 37
  Enrollment: None of the time | 20 | 17
  Enrollment: Less than half the time | 20 | 19
  Enrollment: About half the time | 13 | 9
  Enrollment: More than half of the time | 18 | 22
  Enrollment: All of the time | 27 | 29
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13: Missing | 0 | 1
  Week 13: No sex | 11 | 16
  Week 13: Oral sex only | 10 | 8
  Week 13: No sex with anyone whose HIV status was unknown | 34 | 34
  Week 13: None of the time | 24 | 19
  Week 13: Less than half the time | 9 | 15
  Week 13: About half the time | 10 | 5
  Week 13: More than half of the time | 16 | 19
  Week 13: All of the time | 19 | 22
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26: Missing | 0 | 1
  Week 26: No sex | 18 | 14
  Week 26: Oral sex only | 17 | 9
  Week 26: No sex with anyone whose HIV status was unknown | 28 | 40
  Week 26: None of the time | 14 | 21
  Week 26: Less than half the time | 11 | 13
  Week 26: About half the time | 7 | 6
  Week 26: More than half of the time | 13 | 10
  Week 26: All of the time | 16 | 17
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39: Missing | 0 | 2
  Week 39: No sex | 13 | 13
  Week 39: Oral sex only | 13 | 9
  Week 39: No sex with anyone whose HIV status was unknown | 37 | 50
  Week 39: None of the time | 13 | 10
  Week 39: Less than half the time | 10 | 10
  Week 39: About half the time | 6 | 3
  Week 39: More than half of the time | 9 | 10
  Week 39: All of the time | 13 | 21
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52: Missing | 4 | 6
  Week 52: No sex | 18 | 12
  Week 52: Oral sex only | 2 | 9
  Week 52: No sex with anyone whose HIV status was unknown | 40 | 53
  Week 52: None of the time | 11 | 9
  Week 52: Less than half the time | 8 | 6
  Week 52: About half the time | 5 | 3
  Week 52: More than half of the time | 13 | 4
  Week 52: All of the time | 14 | 18
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65: Missing | 4 | 7
  Week 65: No sex | 16 | 18
  Week 65: Oral sex only | 6 | 2
  Week 65: No sex with anyone whose HIV status was unknown | 42 | 46
  Week 65: None of the time | 16 | 15
  Week 65: Less than half the time | 6 | 3
  Week 65: About half the time | 2 | 6
  Week 65: More than half of the time | 7 | 9
  Week 65: All of the time | 10 | 16
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78: Missing | 9 | 4
  Week 78: No sex | 23 | 20
  Week 78: Oral sex only | 2 | 0
  Week 78: No sex with anyone whose HIV status was unknown | 44 | 53
  Week 78: None of the time | 15 | 15
  Week 78: Less than half the time | 11 | 5
  Week 78: About half the time | 2 | 7
  Week 78: More than half of the time | 9 | 8
  Week 78: All of the time | 10 | 17

17. Secondary Outcome: Examining Changes in Sexual Risk-taking Behavior
Description: Frequency of being high on drugs/drunk during sex, measured by assessments at enrollment and quarterly through Week 78.
Time Frame: 0-18 months
Population: Number of participants who completed CASI questionnaire per visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment: Missing | 0 | 1
  Enrollment: No sex | 9 | 12
  Enrollment: Oral sex only | 10 | 7
  Enrollment: None of the time | 68 | 52
  Enrollment: Less than half the time | 34 | 40
  Enrollment: About half the time | 6 | 13
  Enrollment: More than half of the time | 12 | 15
  Enrollment: All of the time | 7 | 10
  Enrollment: Prefer not to answer | 1 | 3
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13: Missing | 0 | 1
  Week 13: No sex | 11 | 16
  Week 13: Oral sex only | 10 | 8
  Week 13: None of the time | 72 | 53
  Week 13: Less than half the time | 19 | 27
  Week 13: About half the time | 9 | 16
  Week 13: More than half of the time | 4 | 12
  Week 13: All of the time | 7 | 3
  Week 13: Prefer not to answer | 1 | 3
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26: Missing | 0 | 1
  Week 26: No sex | 18 | 14
  Week 26: Oral sex only | 17 | 9
  Week 26: None of the time | 57 | 54
  Week 26: Less than half the time | 21 | 33
  Week 26: About half the time | 2 | 8
  Week 26: More than half of the time | 2 | 6
  Week 26: All of the time | 5 | 6
  Week 26: Prefer not to answer | 2 | 0
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39: Missing | 0 | 2
  Week 39: No sex | 13 | 13
  Week 39: Oral sex only | 13 | 9
  Week 39: None of the time | 51 | 51
  Week 39: Less than half the time | 18 | 28
  Week 39: About half the time | 8 | 11
  Week 39: More than half of the time | 5 | 7
  Week 39: All of the time | 3 | 6
  Week 39: Prefer not to answer | 3 | 1
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52: Missing | 4 | 6
  Week 52: No sex | 18 | 12
  Week 52: Oral sex only | 2 | 9
  Week 52: None of the time | 54 | 47
  Week 52: Less than half the time | 21 | 25
  Week 52: About half the time | 6 | 8
  Week 52: More than half of the time | 3 | 6
  Week 52: All of the time | 4 | 6
  Week 52: Prefer not to answer | 3 | 1
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65: Missing | 4 | 7
  Week 65: No sex | 16 | 18
  Week 65: Oral sex only | 6 | 2
  Week 65: None of the time | 58 | 51
  Week 65: Less than half the time | 15 | 22
  Week 65: About half the time | 5 | 11
  Week 65: More than half of the time | 2 | 3
  Week 65: All of the time | 2 | 4
  Week 65: Prefer not to answer | 1 | 4
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78: Missing | 9 | 4
  Week 78: No sex | 23 | 20
  Week 78: Oral sex only | 2 | 0
  Week 78: None of the time | 57 | 55
  Week 78: Less than half the time | 18 | 29
  Week 78: About half the time | 5 | 11
  Week 78: More than half of the time | 6 | 5
  Week 78: All of the time | 4 | 4
  Week 78: Prefer not to answer | 1 | 1

18. Secondary Outcome: Examining Changes in Sexual Risk-taking Behavior
Description: Had sex for money/drugs/housing/food/other things, measured by assessments at enrollment and quarterly through Week 78.
Time Frame: 0-18 months
Population: Number of participants who completed CASI questionnaire per visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment: Missing | 147 | 153
  Enrollment: No | 0 | 0
  Enrollment: Yes | 0 | 0
  Enrollment: Prefer not to answer | 0 | 0
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13: Missing | 0 | 1
  Week 13: No | 90 | 101
  Week 13: Yes | 40 | 32
  Week 13: Prefer not to answer | 3 | 5
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26: Missing | 0 | 1
  Week 26: No | 85 | 101
  Week 26: Yes | 36 | 24
  Week 26: Prefer not to answer | 3 | 5
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39: Missing | 0 | 0
  Week 39: No | 83 | 104
  Week 39: Yes | 29 | 21
  Week 39: Prefer not to answer | 2 | 3
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52: Missing | 2 | 0
  Week 52: No | 75 | 92
  Week 52: Yes | 37 | 23
  Week 52: Prefer not to answer | 1 | 5
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65: Missing | 0 | 0
  Week 65: No | 77 | 99
  Week 65: Yes | 29 | 21
  Week 65: Prefer not to answer | 3 | 2
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78: Missing | 0 | 0
  Week 78: No | 90 | 107
  Week 78: Yes | 32 | 19
  Week 78: Prefer not to answer | 3 | 3

19. Secondary Outcome: Prevalence of STI Infection (GC, CT, Syphilis) at Baseline
Description: To determine baseline prevalence of STIs (Neisseria gonorrhoeae [GC], Chlamydia trachomatis [CT], and Treponema pallidum (syphilis)) by study arm
Time Frame: 0 months
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Gonorrhea | 15 | 15
  Chlamydia Trachomatis | 15 | 15
  Syphilis (Positive/Reactive) | 38 | 32
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Calculating the odds of Gonorrhea; Test type: Other — The odds ratio was calculated with the deferred intervention arm as the reference group; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.45 to 2.03]
Statistical Analysis 2: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Calculating the odds of Chlamydia Trachomatis; Test type: Other — The odds ratio was calculated with the deferred intervention arm as the reference group; p = 0.91, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.45 to 2.03]
Statistical Analysis 3: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Calculating the odds of a syphilis positive/reactive test; Test type: Other — The odds ratio was calculated with the deferred intervention arm as the reference group; p = 0.32, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.45 to 1.30]

20. Secondary Outcome: Estimate Prevalence of Baseline Laboratory Values.
Description: To obtain baseline laboratory data to evaluate the cohort's suitability for future PrEP intervention studies (e.g., prevalence of renal insufficiency, hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, etc.). Logistic regression models will be used for estimating prevalence of baseline conditions.
Time Frame: 0 months
Population: Enrolled participants. There is insufficient data (below the lower limit of quantification) to perform valid logistic regression modelling on participants with Hepatitis B or renal insufficiency at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Hepatitis B Infection | 0 | 1
  Hepatitis C Infection | 2 | 3
  Renal Insufficiency | 0 | 0
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Logistic regression results of Hepatitis C infection at baseline; Test type: Superiority; p = 0.69, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.24 to 8.81]

21. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Taken hormones for gender identity/transition
Time Frame: 0-18 months
Population: Number of participants who completed the CASI form at each study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment | 96 | 101
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13 | 91 | 96
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26 | 93 | 93
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39 | 85 | 96
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52 | 86 | 93
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65 | 82 | 90
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78 | 93 | 96

22. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Currently taking hormones for gender identity/transition
Time Frame: 0-18 months
Population: Number of participants who completed the CASI form at each study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment | 83 | 90
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13 | 88 | 92
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26 | 89 | 91
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39 | 84 | 90
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52 | 85 | 88
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65 | 79 | 88
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78 | 90 | 91

23. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Where do you currently get your hormones?
Time Frame: 0-18 months
Population: Number of participants who reported they were currently taking hormones.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 83 | 90
  Enrollment: Missing | 0 | 0
  Enrollment: Only from medical providers | 47 | 50
  Enrollment: Medical providers and from friends, online, or other sources | 14 | 11
  Enrollment: Only from friends, online, or other non-licensed sources | 16 | 21
  Enrollment: Some other source | 6 | 8
  Week 13: number analyzed (Participants) | 88 | 92
  Week 13: Missing | 0 | 0
  Week 13: Only from medical providers | 70 | 72
  Week 13: Medical providers and from friends, online, or other sources | 11 | 13
  Week 13: Only from friends, online, or other non-licensed sources | 1 | 3
  Week 13: Some other source | 6 | 4
  Week 26: number analyzed (Participants) | 89 | 91
  Week 26: Missing | 0 | 0
  Week 26: Only from medical providers | 68 | 80
  Week 26: Medical providers and from friends, online, or other sources | 13 | 7
  Week 26: Only from friends, online, or other non-licensed sources | 1 | 4
  Week 26: Some other source | 7 | 0
  Week 39: number analyzed (Participants) | 84 | 90
  Week 39: Missing | 0 | 0
  Week 39: Only from medical providers | 65 | 78
  Week 39: Medical providers and from friends, online, or other sources | 14 | 9
  Week 39: Only from friends, online, or other non-licensed sources | 3 | 0
  Week 39: Some other source | 2 | 3
  Week 52: number analyzed (Participants) | 85 | 88
  Week 52: Missing | 0 | 0
  Week 52: Only from medical providers | 69 | 74
  Week 52: Medical providers and from friends, online, or other sources | 10 | 13
  Week 52: Only from friends, online, or other non-licensed sources | 4 | 1
  Week 52: Some other source | 2 | 0
  Week 65: number analyzed (Participants) | 79 | 88
  Week 65: Missing | 0 | 0
  Week 65: Only from medical providers | 59 | 70
  Week 65: Medical providers and from friends, online, or other sources | 17 | 17
  Week 65: Only from friends, online, or other non-licensed sources | 2 | 1
  Week 65: Some other source | 1 | 0
  Week 78: number analyzed (Participants) | 90 | 91
  Week 78: Missing | 0 | 0
  Week 78: Only from medical providers | 68 | 71
  Week 78: Medical providers and from friends, online, or other sources | 17 | 18
  Week 78: Only from friends, online, or other non-licensed sources | 5 | 2
  Week 78: Some other source | 0 | 0

24. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Ever had a substance (like silicone or other fillers) injected to fill out face or make figure look more womanly
Time Frame: 0-18 months
Population: Number of participants who completed the CASI form at each study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment | 27 | 29
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13 | 2 | 5
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26 | 5 | 4
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39 | 5 | 3
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52 | 6 | 7
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65 | 3 | 3
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78 | 4 | 5

25. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Ever had breast augmentation/surgery
Time Frame: 0-18 months
Population: Number of participants who completed the CASI form at each study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment | 36 | 25
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13 | 3 | 1
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26 | 5 | 1
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39 | 3 | 1
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52 | 5 | 0
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65 | 4 | 0
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78 | 1 | 1

26. Secondary Outcome: Gender-Affirming Hormone Therapy by Visit
Description: Ever had vaginoplasty/labiaplasty/SRS/GRS/GCS
Time Frame: 0-18 months
Population: Number of participants who completed the CASI form at each study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants
  Enrollment: number analyzed (Participants) | 147 | 153
  Enrollment | 7 | 7
  Week 13: number analyzed (Participants) | 133 | 139
  Week 13 | 1 | 0
  Week 26: number analyzed (Participants) | 124 | 131
  Week 26 | 1 | 0
  Week 39: number analyzed (Participants) | 114 | 128
  Week 39 | 1 | 1
  Week 52: number analyzed (Participants) | 115 | 120
  Week 52 | 1 | 0
  Week 65: number analyzed (Participants) | 109 | 122
  Week 65 | 1 | 0
  Week 78: number analyzed (Participants) | 125 | 129
  Week 78 | 2 | 1

27. Secondary Outcome: Annual Incidence of HIV Infections
Description: The number of incident HIV infections at each time point by arm.
  Note: The HIV infection reported at Week 26 occurred during an interim visit between Week 26 and Week 39.
Time Frame: 0-18 months
Population: Enrolled participants
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
participants
  Enrollment | 0 | 0
  Week 13 | 0 | 0
  Week 26 | 1 | 0
  Week 39 | 2 | 1
  Week 52 | 0 | 0
  Week 65 | 0 | 0
  Week 78 | 2 | 0
Statistical Analysis 1: Comparison: Immediate Intervention Arm; Poisson regression models with person time were used to estimate HIV incidence for the immediate intervention arm; Test type: Superiority; Incidence Rate = 1.92, 95% CI 2-sided [0.72 to 5.12]
Statistical Analysis 2: Comparison: Deferred Intervention Arm; Poisson regression models with person time was used to estimate HIV incidence for the deferred intervention arm; Test type: Superiority; Incidence Rate = 0.48, 95% CI 2-sided [0.07 to 3.39]

28. Secondary Outcome: Incidence of STI Infection (GC, CT, Syphilis)
Description: To determine annual incidence of STIs (Neisseria gonorrhoeae [GC], Chlamydia trachomatis [CT], and Treponema pallidum (syphilis)) and to examine changes in STI over time by study arm.
Time Frame: 0-18 months
Population: Enrolled participants
Measure: Number; unit: participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
participants
  Number of STI infections (first incidence) | 51 | 51
  Week 13 | 8 | 21
  Week 26 | 17 | 10
  Week 39 | 4 | 8
  Week 52 | 7 | 1
  Week 65 | 7 | 6
  Week 78 | 8 | 5
Statistical Analysis 1: Comparison: Immediate Intervention Arm; Incidence rate of STIs for immediate intervention arm; Test type: Superiority; p = 0.93, Poisson Regression; Incidence Rate = 31.47, 95% CI 2-sided [23.86 to 41.51] — Incidence Rate of any STI Incidence per Person-Years using Poisson Regression was calculated
Statistical Analysis 2: Comparison: Deferred Intervention Arm; Incidence rate of STIs for deferred intervention arm; Test type: Superiority; p = 0.93, Poisson Regression; Incidence Rate = 32.01, 95% CI 2-sided [23.92 to 42.83] — Incidence Rate of any STI Incidence per Person-Years using Poisson Regression was calculated
Statistical Analysis 3: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Poisson regression was used to compare the incidence rate of STIs by arm; Test type: Superiority; p = 0.93, Poisson Regression; Poisson Regression = 31.74, 95% CI 2-sided [25.96 to 38.80] — Incidence Rate of any STI Incidence per Person-Years using Poisson Regression was calculated

29. Secondary Outcome: Identify Demographic, Behavioral, Socioeconomic, and Psychosocial Factors Related to PrEP Uptake
Description: PrEP uptake is defined as whether the participant initiated PrEP at the study clinic during the study cycle.
Time Frame: 0-18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants | 131 | 137
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable logistic regression modeled PrEP uptake using age, highest level of education, and physical violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 190 of 304). This section presents p-values and odds ratios for age; Test type: Superiority; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.89 to 6.69] — Estimates are for age group 26+ compared to 25 or less
Statistical Analysis 2: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable logistic regression modeled PrEP uptake using age, highest level of education, and physical violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 190 of 304). This section provides p-values and odds ratio estimates for education; Test type: Superiority; p = 0.37, Regression, Logistic; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.05 to 3.16] — Estimates are for comparison of highest level of education primary school vs. college
Statistical Analysis 3: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; [analysis description as in outcome 29, analysis 2]; Test type: Superiority; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.17 to 0.98] — Estimates are for comparison of highest level of education high school vs. college
Statistical Analysis 4: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable logistic regression modeled PrEP uptake using age, highest level of education, and physical violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 190 of 304). This section provides p-values and odds ratio estimates for physical violence; Test type: Superiority; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.98 to 5.28] — Estimates are for comparison of physical violence yes vs. no
Statistical Analysis 5: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable logistic regression modeled PrEP uptake using age, highest level of education, and physical violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 190 of 304).This section provides p-values and odds ratio estimates for physical violence; Test type: Superiority; p = 0.97, Regression, Logistic; Odds Ratio (OR) = 999.99, 95% CI 2-sided [0.001 to 999.99] — Estimates are for comparison of physical violence prefer not answer vs. no (not estimable)

30. Secondary Outcome: Identify Demographic, Behavioral, Socioeconomic, and Psychosocial Factors Associated With PrEP Adherence Across Study Visits.
Description: The number of study visits at which participants were highly adherent to PrEP, among those who initiated PrEP at the study clinic. High adherence at a given visit is determined using drug concentrations in dried blood spots (DBS):
  Truvada: TFV-DP ≥ 900 fmol/punch Descovy: TFV-DP ≥ 950 fmol/punch
  Arm-level results are presented as the total number of visits at which participants in each arm were highly adherent to PrEP, reported as the number and percentage of visits.
Time Frame: 0-18 months
Population: A total of 268 participants initiated PrEP at the study clinic. High PrEP adherence was assessed across 1,533 study visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
Number analyzed (Visits) | 732 | 801
Visits | 291 | 377
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable GEE modeling the probability of high PrEP adherence with predictor emotional violence adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to visits with complete data (1518 of 1533 visits). This section provides p-values and odds ratio estimates for emotional violence; Test type: Superiority; p = 0.8, GEE; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.64 to 1.40] — Estimates are for group emotional violence yes vs. no
Statistical Analysis 2: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; [analysis description as in outcome 30, analysis 1]; Test type: Superiority; p = 0.004, GEE; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.35 to 4.92] — Estimates are for group emotional violence prefer not to answer vs. no

31. Secondary Outcome: Identify Demographic, Behavioral, Socioeconomic, and Psychosocial Factors Related to PrEP Persistence
Description: PrEP persistence is defined as the proportion of study visits at which a participant demonstrates high adherence to PrEP among participants who initiated PrEP at the study clinic. High adherence at a given visit is determined using drug concentrations in dried blood spots (DBS):
  Truvada: TFV-DP ≥ 900 fmol/punch
  Descovy: TFV-DP ≥ 950 fmol/punch
  PrEP persistence reflects sustained high adherence across multiple visits over time per participant, rather than overall high adherence at all time points. For each participant, this proportion was converted to a percentage; arm-level results are presented as the mean of participant-level percentages in each arm in the outcome measure data table.
Time Frame: 0-18 months
Population: Participants who obtained PrEP at the study clinic.
Measure: Mean (Standard Error); unit: Percentage of Visits
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 131 | 137
Percentage of Visits | 41.7 (40.9) | 50.5 (43.2)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable linear regression of PrEP persistence with predictors highest level of education and emotional violence adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 252 of 268). This section provides p-values and odds ratio estimates for highest level of education; Test type: Superiority; p = 0.08, Regression, Linear; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.39 to 0.02] — Estimates are for highest level of education primary school vs. college
Statistical Analysis 2: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable linear regression of PrEP persistence with predictors highest level of education, and emotional violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 252 of 268). This section provides p-values and odds ratio estimates for the highest level of education; Test type: Superiority; p = 0.06, Regression, Linear; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.22 to 0.003] — Estimates are for highest level of education high school vs. college
Statistical Analysis 3: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Multivariable linear regression of PrEP persistence with predictors highest level of education, and emotional violence, adjusting for site. Only predictors significant in univariable analysis were included-study arm was excluded due to lack of significance. Analysis was limited to participants with complete data (N = 252 of 268). This section provides p-values and odds ratio estimates for emotional violence; Test type: Superiority; p = 0.76, Regression, Linear; Mean Difference (Final Values) = -0.016, 95% CI 2-sided [-0.12 to 0.09]; Estimates are for group emotional violence yes vs. no
Statistical Analysis 4: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; [analysis description as in outcome 31, analysis 3]; Test type: Superiority; p = 0.09, Regression, Linear; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-0.06 to 0.78]; Estimates are for group emotional violence prefer not to answer vs. no

32. Secondary Outcome: Identify Demographic, Behavioral, Socioeconomic, and Psychosocial Factors Related to Interest in Future HIV Research
Description: An overall composite flag (Yes/No) for interest in future HIV research was created at the end of study using participant responses collected at enrollment, weeks 26, 52, and 78. Those who showed interest in future HIV research (Yes) were reported in the outcome measure data table.
Time Frame: 0-18 months
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm
Number analyzed (Participants) | 149 | 155
Participants | 149 | 153
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Deferred Intervention Arm; Test type: Other; Multivariable logistic regression was pre-specified but not performed because there were too few participants with the outcome absent (i.e., very few 'No' responses), leading to separation and non-estimable/unstable adjusted effect estimates. Results for "Yes" responses are presented descriptively (counts and percentages) by arm in the outcome measure data table

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up (0-18 months)
Description: Adverse events were reported by intervention. Immediate Arm participants received PrEP, GAHT, and peer-health management from enrollment to study exit. Deferred Arm participants received PrEP throughout, but GAHT and peer-health management only from month 6 onward. Therefore, adverse events for the Deferred Arm were split into 0-6 and 6-18 month periods, using the same denominator for both.
Groups:
- Deferred Intervention Arm (0-6 Months); Deferred Intervention Arm (6-18 Months): PrEP was provided from enrollment to study exit. GAHT and peer-health management were offered from month 6 (week 26) to study exit.
Arm/Group | Immediate Intervention Arm | Deferred Intervention Arm (0-6 Months) | Deferred Intervention Arm (6-18 Months)
All-Cause Mortality (participants affected / at risk) | 2/149 | 0/155 | 0/155
Serious Adverse Events (participants affected / at risk) | 13/149 | 3/155 | 3/155
Other Adverse Events (participants affected / at risk) | 25/149 | 12/155 | 18/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention Arm (N=149) | Deferred Intervention Arm (0-6 Months) (N=155) | Deferred Intervention Arm (6-18 Months) (N=155)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention Arm (N=149) | Deferred Intervention Arm (0-6 Months) (N=155) | Deferred Intervention Arm (6-18 Months) (N=155)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 5 (5) | 3 (3) | 5 (5)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Creatinine renal clearance decreased (Investigations) | 13 (14) | 5 (5) | 13 (15)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04742491/Prot_SAP_ICF_001.pdf